CLINICAL TRIAL: NCT00565734
Title: An Assessment of Surgical Techniques for Treating Cervical Spondylotic Myelopathy
Brief Title: Surgical Treatment of Cervical Spondylotic Myelopathy
Status: Completed | Type: Observational
Sponsor: AO Clinical Investigation and Publishing Documentation (Other)
Collaborators: AO Foundation, AO Spine (Other)
Responsible Party: Sponsor
Organization: AO Innovation Translation Center (Other)
Other Study IDs: CSM-I 07
Record Dates: First submitted 2007-11-29; First posted 2007-11-30 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Cervical Spondylotic Myelopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Posterior surgical approaches: Posterior surgical approaches for symptomatic cervical spondylotic myelopathy (CSM)
- Anterior surgical approaches: Anterior surgical approaches for symptomatic cervical spondylotic myelopathy (CSM).

SUMMARY:
The primary purposes of this study are to compare anterior and posterior surgical approach in treatment of CSM ad to compare variations in treatment and outcomes of CSM worldwide.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Willing and able to give written informed consent to participate in the study
* Willing and able to participate in the study follow-up according to the protocol
* Willing and able to comply with post-operative management program
* Understand and read country language at elementary level
* Patients who undergo surgery for symptomatic CSM defined as a combination of one or more of the following symptoms:
* Numb hands
* Clumsy hands
* Impairment of gait
* Bilateral arm paresthesiae
* l'Hermitte's phenomena
* Weakness

AND one or more of the following signs:

* Corticospinal distribution motor deficits
* Atrophy of hand intrinsic muscles
* Hyperreflexia
* Positive Hoffman sign
* Upgoing plantar responses
* Lower limb spasticity
* Broad based, unstable gait

Exclusion Criteria:

* Asymptomatic CSM
* Previous surgery for CSM
* Active infection
* Neoplastic disease
* Rheumatoid arthritis
* Ankylosing spondylitis
* Trauma
* Concomitant symptomatic lumbar stenosis
* Pregnant women or women planning to get pregnant during the study period
* Has a history of substance abuse (recreational drugs, alcohol)
* Is a prisoner
* Is currently involved in a study with similar purpose
* Has a disease process that would preclude accurate evaluation (eg., neuromuscular disease, significant psychiatric disease)
* Patients seen by other services (eg., physical medicine, neurology, family practice), managed conservatively and not referred for surgical consultation are ineligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic CSM who referred for surgical consultation to the corresponding participating site's orthopedic or neurosurgery services will be eligible for this study.
Sampling Method: Non-Probability Sample
Enrollment: 479 (Actual)
Dates: Start 2007-11; Primary Completion 2014-09 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Surgical complications and neurological, functional, disease-specific and quality of life measures | 24 months

SECONDARY OUTCOMES:
Differences in patient presentation, treatment approaches and treatment outcomes among ethnic/racial groups, health care systems and regions of the world | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Fehlings, MD, PhD, Principal Investigator — University of Troronto
Locations (1):
- Univerity of Toronto, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Bak AB, Moghaddamjou A, Arnold PM, Harrop JS, Fehlings MG. Chronic pain after decompression for degenerative cervical myelopathy: a pooled trajectory analysis of individual participant data. Pain. 2025 Oct 15. doi: 10.1097/j.pain.0000000000003828. Online ahead of print. PMID 41086299
- [Derived] Wong R, Alvi MA, Quddusi AI, Fehlings MG. Role of Neck Pain in Defining Clinical Trajectories of Outcomes in Patients With Degenerative Cervical Myelopathy: Results of a Novel Machine Learning Algorithm. Global Spine J. 2025 May 10;16(1):21925682251341263. doi: 10.1177/21925682251341263. Online ahead of print. PMID 40347099
- [Derived] Pedro KM, Alvi MA, Hejrati N, Moghaddamjou A, Fehlings MG. Elderly Patients Show Substantial Improvement in Health-Related Quality of Life After Surgery for Degenerative Cervical Myelopathy Despite Medical Frailty: An Ambispective Analysis of a Multicenter, International Data Set. Neurosurgery. 2024 Jan 10. doi: 10.1227/neu.0000000000002818. Online ahead of print. PMID 38197642
- [Derived] Merali ZG, Witiw CD, Badhiwala JH, Wilson JR, Fehlings MG. Using a machine learning approach to predict outcome after surgery for degenerative cervical myelopathy. PLoS One. 2019 Apr 4;14(4):e0215133. doi: 10.1371/journal.pone.0215133. eCollection 2019. PMID 30947300